CLINICAL TRIAL: NCT04852601
Title: ToolBox Detect: Low Cost Detection of Cognitive Decline in Primary Care Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: ACCESS Community Health Network (Other)
Responsible Party: Principal Investigator, Michael S. Wolf, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: R01AG069762 (NIH)
Record Dates: First submitted 2021-04-14; First posted 2021-04-21 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Dysfunction; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ToolboxDetect Strategy (Experimental): All practices randomized to the intervention arm will implement the ToolboxDetect battery as the standard of care routine cognitive assessment to fulfill the Medicare Annual Wellness Visit (AWV) requirement. The 7-8 minute ToolboxDetect battery contains self-administered versions of the NIH ToolBox Picture Sequence Memory Test (PSM) and the NIH ToolBox Dimensional Change Card Sorting (DCCS). PSM measures episodic memory and DCCS tests executive functioning.
  The validated ToolboxDetect application will be imparted either as an application on an iPad or on a PC desktop/laptop computer commonly found in a clinical exam room for EHR access.
  Interventions: Other: ToolboxDetect
- Enhanced Usual Care (No Intervention): At Northwestern Medicine, cognitive assessments included in Annual Wellness Visits or other routine or sick/problem-based visits vary by practice and also by clinician. However, the choice of test was limited to either a Mini-Cog©, Montreal Cognitive Assessment (MoCA), or Mini Mental Status Exam (MMSE).
  While we will not make any explicit recommendations to these practices with regard to their use of a cognitive assessment, we will ensure that 1) any chosen test is linked to an Epic SmartData element, which will allow the clinician to record the results of the test as discrete data (which can then be queried), and that 2) providers receive a compiled list of local medical and non-medical referrals for any detected cases of CI. The Alzheimer's Association recommendations for early detection efforts among primary care practices will also be provided to each clinic's medical leadership.

INTERVENTIONS:
Other: ToolboxDetect — The clinician or staff member will identify the patient by either scanning a barcode or entering his/her name, age and medical record number on an administrative screen (allowing for proper routing of test results). After completing the test, a 'submit' button will automatically generate a secure HL7 message, sharing 1) a binary classification of the results ('impaired cognition' or 'normal function'), 2) the quantitative ToolboxDetect score, and 3) brief clinical decision support to rule out any reversible causes. These results will be linked to a discrete, queriable, Epic SmartData element. As patients undergo multiple AWVs over time, ToolboxDetect quantitative scores will be displayed in Epic Synopsis Activity, a graphical display that can visualize trend data (e.g. patient vitals) and calculate a percentage change from the prior year. This will allow a clinician to establish a patient's own baseline (instead of using normative data only) for reference.
  Arms: ToolboxDetect Strategy

SUMMARY:
Our study objective is to widely implement and evaluate a user-centered, scalable, electronic health record (EHR)-linked strategy for the routine detection of cognitive decline among diverse primary care settings. This strategy, called ToolboxDetect, will provide an efficient and sensitive cognitive screen that can be easily implemented in everyday clinical settings, and is responsive to patient, family, and caregiver concerns for potential symptoms of cognitive decline (CD) and cognitive impairment (CI).

DETAILED DESCRIPTION:
Our study objective is to widely implement and evaluate a user-centered, scalable, electronic health record (EHR)-linked strategy for the routine detection of cognitive decline among diverse primary care settings. We will conduct a large-scale, primary care practice-randomized trial to implement and comprehensively evaluate ToolboxDetect as a standard of care with AWVs, linked to an EHR (Epic). Diverse, academic and community settings are included to optimize future dissemination efforts.

ToolboxDetect is an iPad-based, self-administered assessment that leverages two well validated measures from the NIH Toolbox Cognition Battery: Dimensional Change Card Sorting (for executive function) and the Picture Sequence Memory (for episodic memory). It takes approximately 7-8 minutes to administer, and for practices randomized to the ToolboxDetect arm, this will be used as the practice standard to fulfill the requirement for cognitive testing as part of the Medicare Annual Wellness Visit (AWV).

The aims of our investigation are to:

1. Evaluate the effectiveness of ToolboxDetect, compared to enhanced usual care, to promote timely detection of cognitive decline and its care management.
2. Disseminate and implement ToolboxDetect among a large Federally Qualified Health Center Network and assess its feasibility and acceptability for use;
3. Investigate the fidelity of ToolboxDetect, and identify any patient, caregiver, healthcare provider and/or system barriers to its optimal, sustained implementation;
4. Determine costs associated with implementing ToolboxDetect from a primary care perspective.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 65 and older will be considered.
2. Adults who may or may not have cognitive impairments.
3. Practices affiliated with Northwestern Medicine and Access Community Health Network.

Exclusion Criteria:

1. Severe, uncorrectable vision or hearing impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41500 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of detected impairment | Up to 3 years
  This will be operationalized as either results of an any administered cognitive test suggesting impairment ('detected'), or having any relevant ICD 10 classification code recorded in a patient's record after the trial launch date and throughout follow-up observation period ('diagnosis').

SECONDARY OUTCOMES:
Rate of cognitive testing | Up to 3 years
  Extraction from the enterprise data warehouse (EDW) of elements used to document cognitive assessment
Rate of detected cases with mild impairment | Up to 3 years
  Mild vs. other impairment rates will be compared across trial arms, operationalized by ICD code groupings.
Rate of cognition-related referrals | Up to 3 years
  Extraction from the electronic data warehouse for whether or not a cognitive-related referral was made (medical or non-medical) following a "detected" cognitive screen
Caregiver involvement | Up to 3 years
  Text search of clinic note from any follow-up visit post AWV, wellness visit mention of accompanying family member/caregiver; extraction from EDW to determine if proxy access to patient's MyChart portal has been shared.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No